CLINICAL TRIAL: NCT06154304
Title: To Compare the Bronchoprotective Effects of the Test and Reference Metered Dose Inhalers (MDIs) Containing Albuterol Sulfate Using Methacholine Bronchoprovocation Challenge Testing in Stable Mild Asthma Patients.
Brief Title: BE Study of Albuterol Sulfate Inhalation Aerosol 90 mcg Per Actuation in Patients With Stable Mild Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cipla Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CRD/58
Record Dates: First submitted 2023-11-23; First posted 2023-12-04 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo Product (Placebo Comparator): One actuation each from four different placebo inhalation aerosols.
  Interventions: Drug: Placebo
- Test Product (Experimental): One actuation from the test inhalation aerosol and one actuation each from three different placebo inhalation aerosols
  Interventions: Drug: Albuterol Sulfate Inhalation Aerosol (90 mcg per actuation)
- Reference 90mcg Product (Active Comparator): One actuation from the reference inhalation aerosol and one actuation each from three different placebo inhalation aerosols.
  Interventions: Drug: Ventolin HFA 90Mcg/Actuation Inhalation Aerosol_#1
- Reference 180mcg Product (Active Comparator): One actuation each from two different reference inhalation aerosols and one actuation each from two different placebo inhalation aerosols
  Interventions: Drug: Ventolin HFA, 90 Mcg/Inh Inhalation Aerosol_#2

INTERVENTIONS:
Drug: Albuterol Sulfate Inhalation Aerosol (90 mcg per actuation) — 90 mcg
  Other Names: Albuterol Test Product
  Arms: Test Product
Drug: Ventolin HFA 90Mcg/Actuation Inhalation Aerosol_#1 — 90 mcg
  Other Names: Albuterol Reference Product
  Arms: Reference 90mcg Product
Drug: Ventolin HFA, 90 Mcg/Inh Inhalation Aerosol_#2 — 180 mcg
  Other Names: Albuterol Reference Product
  Arms: Reference 180mcg Product
Drug: Placebo — Placebo
  Arms: Placebo Product

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product, using bronchoprovocation (methacholine challenge testing) in adult patients with stable mild asthma.

DETAILED DESCRIPTION:
This study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product in terms of FEV1 measured at different time-points, using bronchoprovocation (methacholine challenge testing) in adult patients with stable mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a ≥6-months diagnosis of stable mild asthma based on National Asthma Education and Prevention Program Expert Panel Report 3 (NAEPP EPR3) guidelines (NAEPP EPR3, 2007)
2. Subject must demonstrate an FEV1 ≥1.5L and ≥80% of predicted based on NHANES III predicted values at the pre-challenge/Pre-saline stage of the first screening MBPC

   a. If a subject's FEV1 at the pre-challenge (baseline/Pre-saline) spirometry is <80%, but ≥70%, the screening visit may be rescheduled one time (visit must take place within 7 days)
3. Subject must demonstrate airway responsiveness to methacholine at baseline (pre-albuterol dose) PC20 at ≤8 mg/mL concentration of methacholine (Equivalent to PD20 of ≤513 µg) at the first screening MBPC
4. Subject must have a BMI of ≥18 kg/m2 and ≤35 kg/m2 at screening.

Exclusion Criteria:

1. Subject has a fall in FEV1 at the saline stage ≥10% at the screening MBPC. 2. Subject having FEV1 of less than 1.5L at pre-challenge or saline stage of MBPC at any visit. No re-screening/re-scheduling is allowed for such subjects.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
Provocative Dose of Methacholine Causing 20 % Fall (PD20) in FEV1(Forced Expiratory Volume in 1 second) | 1 day
  • To compare the bronchoprotective effects of the test product, Albuterol Sulfate Inhalation Aerosol (90 mcg per actuation) [InvaGen Pharmaceuticals Inc., (a subsidiary of Cipla Ltd.) Fall River - MA02720] with the Reference product, Ventolin HFA (Albuterol sulfate inhalation aerosol) 90 mcg per actuation (GlaxoSmithKline, USA), as assessed by methacholine bronchoprovocation challenge (MBPC) testing

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Smiley, Principal Investigator — Velocity Clinical Research
Locations (1):
- Velocity CLinical Research, Medford, Oregon, United States

IPD SHARING:
Plan to Share IPD: No